CLINICAL TRIAL: NCT01666210
Title: A Prospective, Multicenter, Randomized, Parallel-Arm, Double-Masked, Vehicle Controlled Phase II Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Ocular Inflammation and Pain After Cataract Surgery
Brief Title: Phase II Study Evaluating Safety/Efficacy of OTX-DP for Treatment of Ocular Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-12-002
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Ocular Inflammation and Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone Punctum Plug (Active Comparator): Sustained and tapered release of dexamethasone from hydrogel punctum plug following insertion over 30 days
  Interventions: Drug: OTX-DP (Dexamethasone punctum plug)
- Placebo Vehicle Punctum Plug (Placebo Comparator): Placebo punctum plug insertion
  Interventions: Drug: Placebo Vehicle Punctum Plug

INTERVENTIONS:
Drug: OTX-DP (Dexamethasone punctum plug) — Sustained and tapered release of dexamethasone from hydrogel punctum plug
  Arms: Dexamethasone Punctum Plug
Drug: Placebo Vehicle Punctum Plug — Hydrogel punctum plug without dexamethasone
  Arms: Placebo Vehicle Punctum Plug

SUMMARY:
To evaluate the safety and efficacy of OTX-DP as a sustained release drug (dexamethasone) depot when placed in the canaliculus of the eyelid for the treatment of ocular inflammation and pain in subjects who have undergone cataract extraction with intra-ocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent, approved by the appropriate institutional review board; and is able to comply with study requirements and visit schedule
* Is greater than or equal to 21 years of age
* Has a cataract and is expected to undergo clear corneal cataract surgery with phacoemulsification and implantation of a posterior chamber intraocular lens

Exclusion Criteria:

* Any intraocular inflammation in the study eye present during the screening slit lamp examination
* Score greater than "0" on the Ocular Pain Assessment at Screening
* Compromised immune system or an autoimmune disease that in the opinion of the Investigator could affect the quality of the ocular surface

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  Age between 21 - 65 | 14 | 9 | 23
  Age greater than or equal to 65 | 16 | 21 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Absence of Cells in Anterior Chamber of Study Eye
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Number analyzed (Participants) | 30 | 30
Participants | 6 | 3

2. Primary Outcome: Absence of Pain in the Study Eye
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Number analyzed (Participants) | 29 | 30
Participants | 23 | 9

3. Other Pre Specified Outcome: Adverse Events
Description: Measure of adverse events over the duration of each subject's participation in the study.
Time Frame: Duration of each individual subject's participation in the study, up to 60 days
Population: Ocular adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Number analyzed (Participants) | 29 | 30
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: The analyses of safety were based primarily on the incidence of treatment-emergent adverse events up to 60 days.
Description: The number of subjects in the OTX-DP group is confirmed as 29, one subject was not treated due to the inability to insert the plug in either eye.
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/30
Other Adverse Events (participants affected / at risk) | 3/29 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Punctum Plug (N=29) | Placebo Vehicle Punctum Plug (N=30)
Syncope (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Punctum Plug (N=29) | Placebo Vehicle Punctum Plug (N=30)
Eye disorders (Eye disorders) | 3 (6) | 10 (15) — Visual Acuity Reduced, Conjunctival Hyperemia, Corneal Edema, Anterior Chamber Inflammation, Conjunctival Hemorrhage, Cystoid Macular Edema, Eye Discharge, Eye Disorder, Eye Pain, Iritis, Lenticular Opacities, Photophobia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agree that the first publication of the data and results of the Study shall be made in conjunction with the presentation of a joint, multi-center publication of the Study results, with the investigators from all appropriate sites contributing data, analyses, and comments.